CLINICAL TRIAL: NCT05307029
Title: Immediate Fixed Full-arch Rehabilitation of Edentulous Jaws on 4 or 6 Implants According to the Nobelguide® Protocol: a Retrospective Study on Clinical and Radiographic Outcomes up to 10 Years of Follow-up.
Brief Title: Immediate and Flapless Full-arch Rehabilitation of Edentulous Jaws
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maria Paola Cristalli, DDS PhD, Associate Professor, University of Roma La Sapienza
Other Study IDs: 0000505/26.04.2021
Record Dates: First submitted 2022-01-17; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Edentulous Patients
Keywords: full- arch implant prosthesis; flapless implant surgery; immediate Dental Implant Loading; Surgery; Computer-Assisted; Dental Implants; template-guided surgery; all on four; all on six; ; tilted implants
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A edentulous patients: edentulous patients rehabilitated with fixed full-arch prosthesis on 4 implants
  Interventions: Procedure: rehabilitation with fixed full-arch prosthesis
- Group B edentulous patients: edentulous patients rehabilitated with fixed full-arch prosthesis on 6 implants
  Interventions: Procedure: rehabilitation with fixed full-arch prosthesis

INTERVENTIONS:
Procedure: rehabilitation with fixed full-arch prosthesis

SUMMARY:
The study involved 28 edentulous patients (20 female/8 males; average age of 67.75± 8.627 years) rehabilitated with 33 prostheses (17 all-on-4/16 all-on-6) supported by 164 implants.

DETAILED DESCRIPTION:
Clinical and radiographic outcomes were implants survival, prostheses success/survival, implant marginal bone loss, incidence of biological and prosthetic complications.

ELIGIBILITY:
Inclusion Criteria

* Mandibles or maxillae edentulous or with hopeless teeth;
* Patient's request of fixed implant restorations
* Patients in general good health (ASA-1/ASA-2)

Exclusion Criteria

* Compromised systemic conditions;
* Head/neck irradiation or chemotherapy within 2 years;
* Bisphosphonate therapy;
* Metabolic bone diseases;
* Insufficient bone volume;
* Mouth opening less than 50 mm inadequate to place surgical instrumentations.
* History of periodontitis or smoking habit were not considered exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this retrospective cohort study, participants were recruited from edentulous patients rehabilitated with fixed full-arch prosthesis on 4 or 6 implants according to the Nobelguide® protocol between Jun 2009 and December 2019 at the Oral Surgery Unit, Policlinico Umberto I, "Sapienza" University of Rome, Italy. No randomization was applied.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-02-20 (Actual); Primary Completion 2014-02-10 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Implant marginal bone loss (MBL) | from the functional loading time with the provisional prosthesis (baseline) T0 to the end of the follow-up, assessed up to 10 years and measured in millimeters on periapical radiographs taken every year using the parallel long-cone technique.
  difference in marginal bone level from the functional loading time with the provisional prosthesis (baseline) to the end of the follow-up measured in millimeters/years on periapical radiographs. Periapical radiographs of each implant were taken every year using the parallel long-cone technique and a standardized film holder (Rinn Centratore XCP Evolution 2003, Dentsply, Rome, Italy).
Prosthetic complications | Every 6 months from the functional loading time with the provisional prosthesis (baseline) to the end of the follow-up, assessed up to 10 years.
  included detachment/incisal and occlusal wear/fracture/chipping/replacing of denture teeth, fracture of implant, prosthesis or framework, loosening/fracture of abutment or occlusal screw, loosening/fracture of the prosthetic screw
Biologic complications | Every 6 months from the functional loading time with the provisional prosthesis (baseline) to the end of the follow-up, assessed up to 10 years.
  inflammation / infection under fixed prosthesis, soft tissue hypertrophy / hyperplasia, soft tissue recession / dehiscence, peri-implant mucositis, peri-implantitis.
  Modified plaque index (mPI), modified gingival index (mGI), bleeding on probing (BoP), and probing depth (PD). mPI, mGI, BoP, and PD measurements were performed at 6 aspects per implant. mPI was scored as: 0 = no detection of plaque; 1 = plaque only recognized by running a probe across the smooth marginal surface of the implant; 2 = plaque can be seen by the naked eye; 3 = abundance of soft matter. mGI was scored as: 0 = no bleeding when a periodontal probe is passed along the mucosal margin adjacent to the implant; 1 = isolated bleeding spots visible; 2 = blood forms a confluent red line on mucosal margin; 3 = heavy or profuse bleeding. BoP was scored as 0 = absence; 1 = presence; PD was measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Paola Cristalli, DDS, Study Director — Sapienza University of Roma